CLINICAL TRIAL: NCT01759381
Title: The Efficacy of Negative Pressure Wound Therapy (NPWT) in the Postoperative Management of Complex Spinal Surgeries: A Randomized Outcomes Study.
Brief Title: Incisional Negative Pressure Wound Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00040054
Record Dates: First submitted 2012-12-07; First posted 2013-01-03 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Deformity
Keywords: Spinal Deformity; Complex Spinal Surgery; Negative Pressure Wound Therapy; Post-Operative Infection
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Negative Pressure Wound Therapy Device (No Intervention): This control group will not receive the negative pressure wound therapy device. Post operative dressings will be per the surgeon's standard routine.
- NPWT Arm Therapy (Experimental): This group will receive NPWT as opposed to the standard incisional dressing following complex spinal surgery.
  Interventions: Device: Negative pressure wound therapy (NPWT)

INTERVENTIONS:
Device: Negative pressure wound therapy (NPWT)
  Arms: NPWT Arm Therapy

SUMMARY:
The purpose of this study is to evaluate the outcome of incisional negative pressure wound therapy in preventing surgical site infections and wound complications (dehiscence) in high-risk patients undergoing complex spinal surgery.

DETAILED DESCRIPTION:
This randomized, controlled study will compare the outcomes of NPWT versus the outcomes of not using NPWT in post-operative wound management following a complex spinal surgery. The allocation of patients (no NPWT device versus applying an NPWT device) will be determined by computer-generated randomization. The following data will be collected to determine impact on the outcome of wound management (i.e., infection and wound dehiscence): age, gender, body mass index (BMI), dorsal fat, estimated blood loss during the surgical procedure, length of surgery, length of hospital stay, highest peri-operative glucose, medical comorbidities, and history of infection.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age
* >/= 3 level instrumented thoracic, lumbar, or thoracolumbar spinal fusion

Exclusion Criteria:

* < 18 years of age
* < 3 level instrumented thoracic, lumbar, or thoracolumbar spinal fusion
* Spinal infection at time of surgery
* History of immunosuppression or chronic systemic infection
* Pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Bagley, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NPWT Arm Therapy: This group will receive NPWT as opposed to the standard incisional dressing following complex spinal surgery.
  Negative pressure wound therapy (NPWT)
Period: Overall Study
Arm/Group | No Negative Pressure Wound Therapy Device | NPWT Arm Therapy
Started | 8 | 11
Completed | 7 | 11
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Negative Pressure Wound Therapy Device | NPWT Arm Therapy | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 13
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Post-operative Infection (NPWT)
Description: The patient will be assessed for signs/symptoms of infection within the 3 month post-operative period.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | No Negative Pressure Wound Therapy Device | NPWT Arm Therapy
Number analyzed (Participants) | 7 | 11
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: pre-op - 3 months
Arm/Group | No Negative Pressure Wound Therapy Device | NPWT Arm Therapy
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Negative Pressure Wound Therapy Device (N=8) | NPWT Arm Therapy (N=11)
Death (Nervous system disorders) | 1 (1) | 0 (0) — Patient developed a neurodegenerative disorder while an inpatient, and subsequently passed away. She did not receive the negative pressure wound therapy device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes